CLINICAL TRIAL: NCT02544087
Title: Heat-clearing and Blood-activating Chinese Medicinal Components in Acute Cerebral Infarction: Mechanisms of Multi-target Anti-inflammatory Action
Brief Title: Heat-clearing and Blood-activating Chinese Medicinal Components in Acute Cerebral Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yunling Zhang (Other)
Collaborators: Shandong University of Traditional Chinese Medicine (Other); Huairou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Yunling Zhang, President of Dongfang Hospital, Dongfang Hospital Beijing University of Chinese Medicine
Organization: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2015DFA31130
Record Dates: First submitted 2015-09-05; First posted 2015-09-09 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Ischemic Stroke
Keywords: fire-heat syndrome; blood stasis syndrome; method of clearing heat; method of promoting blood circulation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- The basic treatment (No Intervention): Comply to the Chinese guidlines of acute ischemic stroke in 2014
- Clearing heat (Other): Treat with KDZ injection on the basis of basic treatment
  Interventions: Drug: Ixeris of sonchifolia Hance
- Promoting blood circulaton (Other): Treat with Xueshuantong injection on the basis of basic treatment
  Interventions: Drug: Panax notoginseng saponins
- Clearing heat&Promoting blood circulaton (Experimental): Treat with both KDZ injection and Xueshuantong injection on the basis of basic treatment
  Interventions: Drug: Ixeris of sonchifolia Hance combined with Panax notoginseng saponins

INTERVENTIONS:
Drug: Ixeris of sonchifolia Hance — KDZ40ml+0.9%N.S.250ml,ivdrip,qd of each 14-day cycle.Number of cycles:one.
  Other Names: KDZ injection
  Arms: Clearing heat
Drug: Panax notoginseng saponins — Xueshuantong450mg+0.9%N.S.250ml,ivdrip,qd of each 14-day cycle.Number of cycles:one.
  Other Names: Xueshuantong injections
  Arms: Promoting blood circulaton
Drug: Ixeris of sonchifolia Hance combined with Panax notoginseng saponins — KDZ40ml+0.9%N.S.250ml,ivdrip;Xueshuantong450mg+0.9%N.S.250ml,ivdrip,qd of each 14-day cycle.Number of cycles:one.
  Arms: Clearing heat&Promoting blood circulaton

SUMMARY:
The present study is designed to confirm the therapeutic effects of heat-clearing and blood-activating Chinese medicinal components in treatment of Acute Cerebral Infarction (ACI) and to investigate the therapeutic mechanisms of multi-target anti-inflammatory action involved from the standpoint of pathology, cell and molecular biology, as well as immunology.

DETAILED DESCRIPTION:
The present study is designed to confirm the therapeutic effects of heat-clearing and blood-activating Chinese medicinal components in treatment of Acute Cerebral Infarction (ACI) and to investigate the therapeutic mechanisms of multi-target anti-inflammatory action involved from the standpoint of pathology, cell and molecular biology, as well as immunology. In particular, investigators choose heat-clearing Ixeris of sonchifolia Hance(Kudiezi Injection) and blood-activating Panax notoginseng saponins(Xueshuantong Injection)as the therapeutic interventions to carry out the investigation, applying the key techniques such as Lentivirus-mediated RNA interference, co-immunoprecipitation and immunomagnetic beads.

With the joint efforts, investigators hope to find out the combined therapeutic targets based on better understanding of the inflammatory pathology in ACI and illuminate the synergistic mechanisms involved, which may validate the Chinese medicine theory of"cerebral vascular damage due to heat toxicity" in the pathogenesis of ACI and yield new therapeutic strategies for ACI. As an international science and technology cooperation project, the study is of great significance in establishing an international technology platform of intervention target system for the treatment of ACI; moreover, it marks a key step forward for China to enhance China's international brands through exploring a successful mode of foreign cooperation in Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke
* Patients with fire-heat syndrome
* Stroke onset within 48 hours
* NIHSS scores range from 5 points to 25 points
* Age from forty to eighty,gender not limited
* Informed and signed the consent

Exclusion Criteria:

* Cardiogenic cerebral embolism,stroke caused by other reasons or the unexplained
* Patients suitable for thrombolytic therapy(rt-PA,urokinase),or have recieved thrombolytic therapy
* Patients suitable for endovascular therapy,or have recieved endovascular therapy
* Patients with serious disease of heart,lungs,liver or kidneys（The value of ALT or AST is more than 2 times of the upper limit of normal range,the value of creatinine is more than 1.5 times of the upper limit of normal range，asthma or COPD,or cardiac function level 4）
* Patients with bleeding or bleeding tendency recently
* Pregnant or lactating women
* Pre-existing limb dysfunction, psychiatric diaseses，or cognitive dysfunction that could confound the study results
* Patients with allergic constitutions,or have the contraindication of Ixeris of sonchifolia Hance components(KDZ injection) or Panax notoginseng saponins components(Xueshuantong injection)
* Patients have participated in other clinical trials within 3 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
modified Rankin scale | 180 days

SECONDARY OUTCOMES:
Barthel index | 180 days
national institute of health stroke scale | 180 days
Glasgow coma scale | 180 days
scores of Chinese medicine symptoms | 180 days
mortality rate | 180 days
disability rate | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Yunling Zhang, PhD,MD, Study Chair — Dongfang Hospital Beijing University of Chinese Medicine
Locations (4):
- China (4):
  - Department of Neurology,Dongfang Hospital, Beijing, Beijing Municipality
  - Department of Neurology,Huairou Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Department of Neurology,Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Department of Neurology,Wuqing Hospital of Traditional Chinese Medicine, Tianjin, Tianjin Municipality